CLINICAL TRIAL: NCT07401576
Title: Effects Of Stabilization Exercises On Head Posture, Vocal Efficiency And Pain In Patients With Nonspecific Chronic Neck Pain
Brief Title: Stabilization Training, Voice And Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Dr. Emine Metin, phd, Doctor Physical Therapist, Suleyman Demirel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SuleymanDU1
Record Dates: First submitted 2026-01-08; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neck Pain; Voice Change
Keywords: Vocal Efficiency, Neck Pain and Postural Stability
MeSH Terms: conditions — Neck Pain; Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The purpose of this study is to investigate the effects of cervical stabilization exercises applied (Experimental): The purpose of this study is to investigate the effects of cervical stabilization exercises applied to patients with nonspecific chronic neck pain, the patients' cervical postural alignment, and changes in neck pain-related clinical parameters on voicing efficiency in patients with nonspecific chronic neck pain (NSCNP).
  Interventions: Other: cervical stabilization exercises applied

INTERVENTIONS:
Other: cervical stabilization exercises applied — Head posture (craniocervical angle), pain (VAS, NDI) and vocal efficiency (acoustic analysis, maximum phonation time, VHI) were measured at baseline and completion. Participants were assigned to either a stabilization exercise group or a control group receiving conventional exercises. Outcome measures included Demographics and Clinical Characteristics, head and cervical posture, pain and disability indices, and voicing efficiency parameters such as maximum phonation time (MPT) and s/z ratio. Acoustic voice measures and self-reported voice handicap (Voice Handicap Index, VHI) were also assessed.These assessments were performed twice, before and after treatment. Patients with cronic neck pain were randomly divided into two groups: the Cervical Stabilization Exercise Group (n = 20, male:3, female:17) and the Traditional Exercise Group (n = 18, male:4, female:14). The both group received a total of 24 sessions of an exercise program over a six-week period, with five sessions per week for t
  Other Names: Traditional Exercise , hot pack applied, tens applied

SUMMARY:
This randomized controlled trial investigated the effects of cervical stabilization exercises on head posture, pain, functional status, and voicing efficiency in patients with nonspecific chronic neck pain. Following a six-week exercise program, cervical stabilization exercises resulted in significantly greater improvements in pain intensity, functional disability, craniocervical angle, and maximum phonation time compared with traditional exercises. Both exercise interventions led to significant reductions in pain and improvements in cervical posture; however, no significant changes were observed in acoustic voice parameters. Overall, cervical stabilization exercises demonstrated superior benefits in postural alignment, pain reduction, and functional outcomes.

DETAILED DESCRIPTION:
Neck pain is among the most common musculoskeletal disorders, affecting approximately 20% of adults worldwide (1). Although some cases of acute neck pain resolve spontaneously, approximately half of all cases persist for more than three months, becoming chronic. Efficient and cost effective treatment are needed for the management of non-specific chronic neck pain (NSCNP) in order to decrease the social dens of disability; however, the use of interventions with demonstrated efficacy for specific outcomes is necessary The psychological, physical, and socioeconomic effects of neck pain are of significant importance(2). The majority of neck pain is not due to organic pathology and is therefore classified as "non-specific" or "mechanical."(3) Non-specific chronic neck pain accounts for approximately 20% of outpatient physical therapy visits, and its annual prevalence varies between 27% and 48% in developed countries (4).

Regional neck pain causes a forward tilt of the head, which alters the biomechanics of the cervical vertebrae, and increases the load on the posterior structures of the cervical region, including bones, muscles, ligaments, and the joint capsule. Disruption of vertebral joint biomechanics in the cervical and thoracic regions due to various reasons can cause changes along the kinetic chain. These changes increase the load and stress on the joints and negatively affect the structures around the neck (5). The forward posture of the head is characterized by flexion of the upper thoracic and lower cervical vertebrae, occiput extension on the first cervical vertebra, and increased extension of the upper cervical vertebrae(6) . The forward head posture results in the neck extensors becoming weaker and the front and shoulder muscles of the cervical region becoming shorter. This increases the load on the structures around the shoulder and cervical region due to the effect of gravity. Furthermore, the muscle structures around the shoulder joint and scapula are also affected, thus increasing the prevalence of posture disorders. Secondarily, increased thoracic kyphosis, increased internal rotation of the glenohumeral joint, and weakening of the scapula medial rotation and scapula retractors are observed. Dorsal kyphosis in the upper thoracic spine and medial rotation of the scapula cause a decrease in lung vital capacity with vertical loading. The forward head posture of individuals with non-specific chronic neck pain is more pronounced when standing compared to individuals without neck pain(7) .

Neck pain and associated posture problems also affect respiratory and phonatory mechanisms. Posture problems associated with chronic neck pain result in dysfunctions of the soft tissue and muscle structures around the pharynx and larynx, which have an impact on people's voice control and resonance. The functions of the muscles surrounding the larynx are directly affected by the movements of the cervical vertebrae and cricoid cartilage. Forward head posture (FHP) directly affects not only the neck and shoulder muscles but also the muscles surrounding the larynx (extrinsic and suprahyoid In the FHP model, the geniohyoid and mylohyoid muscles are observed to be particularly stretched, with the possibility of overactivation in the digastric posterior belly and stylohyoid muscles.(Digastricus (anterior and posterior )mylohyoid,geniohyoid, stylohyoid, sternohyoid, infrahyoid, sternothyroid, thyrohyoid, omohyoid) It has the function of retracting the larynx and thereby providing stabilisation. This can alter both the position of the larynx and the muscle activity used during phonation, Furthermore, the coordination of the muscles that form the structure of the neck affects the function of the vocal folds and the position of the hyoid bone. When the head is positioned forward, the muscles under the hyoid bone lengthen, pulling the cervical vertebrae downwards and backwards. This force is transmitted to the lower jaw bone through the muscles above the hyoid bone, causing the tongue to assume a tense position, which affects vocalization. This mechanism increases the mechanical load on the vocal folds during phonation. Any disorder or imbalance in these structures alters the position and tension of the laryngeal muscles and vocal folds, resulting in vocal imbalance and deterioration in voicing efficiency (8, 9). The larynx acts as an energy transducer, converting the Voice Efficiency energy generated by the lungs into the acoustic energy perceived by listeners. This provides an estimate of respiratory-laryngeal coordination.

Physiotherapy and rehabilitation practices are frequently employed as treatment methods for patients with chronic neck pain. Exercise training represents one of the primary physiotherapy methods and is utilized with considerable frequency in treatment. Studies have demonstrated that the incorporation of craniocervical flexion exercises, endurance exercises, aerobic exercises, proprioceptive exercises, and patient education in the treatment of chronic neck pain, particularly in conjunction with cervical stabilization exercises, results in a reduction of pain and an improvement in quality of life, as evidenced by an increase in muscle strength and functions. A stabilisation exercise is a form of intervention that is designed with the objective of protecting and preventing the spinal segment from re-injury. This is achieved by restoring and improving muscle control, thereby compensating for any loss of muscle action that may have been caused by injury or degenerative changes(10, 11) Neck stabilisation exercises are designed to rectify muscle abnormalities and restore the correct function of muscles in order to support and stabilise the spine (12).

Although research on the effectiveness of cervical stabilization exercises for voicing efficiency is scarce, stabilization exercises are recommended in conjunction with voice therapy in patients prone to vocal efficient. It was hypothesized that reducing pain and improving posture by increasing postural awareness along with cervical region stabilization exercises may change the hyoid position, affecting the vocal tract, voice resonance, and voice parameters. Therefore, this study was designed to demonstrate the effects of cervical stabilization exercises, which have been proven effective in treating neck pain and related posture problems, pain and on the phonatory mechanism and voicing efficiency.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-60 years, experiencing nonspecific neck pain for at least three months, and reporting a pain score of ≥3 on a 0-10-cm visual analogue scale (VAS) at rest. Participants also had to volunteer to participate.

Exclusion Criteria:

Previous musculoskeletal injuries of the neck or shoulder; neurological, orthopedic, oncologic, or congenital musculoskeletal disorders; hearing impairment requiring aids; history of head, neck, or laryngeal surgery; recent upper respiratory infection; laryngeal lesions observed on examination; history of voice therapy; severe respiratory dysfunction in the past five years; physical therapy for neck pain within the last six months; tracheobronchial infection during the study period; and pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 10 months
  Visual Analog Scale (VAS)
Vocal Efficiency | 10 months
  Maximum Phonation Time (MPT)
  s/z Ratio

SECONDARY OUTCOMES:
Neck Disability | 10 months
  Neck Disability Index (NDI)
Acoustic Voice Parameters | 10 months
  Fundamental frequency (F0)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdi Ferdi Baskurt, professor, Study Director — Suleyman Demirel University; Emine Metin, phd, Principal Investigator — Suleyman Demirel University
Locations (2):
- Turkey (Türkiye) (2):
  - Suleyman Demirel University Hospital, Isparta
  - Suleyman Demirel University, Isparta

IPD SHARING:
Plan to Share IPD: Yes
I can share it with other researchers if they want.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: sdu